CLINICAL TRIAL: NCT05127213
Title: Comparison of the Effects of Brain Function Changes on Body Weight After Intragastric Balloon Surgery and Sleeve Gastric Surgery
Brief Title: Effects of Intragastric Balloon Surgery and Sleeve Gastrectomy on Brain Function
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XY3-IGBWLG001
Record Dates: First submitted 2021-11-10; First posted 2021-11-19 (Actual); Last update posted 2021-11-19 (Actual); Status verified 2021-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intragastric balloon system group (Experimental): Operation way: intragastric balloon system
  Using the intragastric balloon system to treat obesity.
  Interventions: Procedure: Intragastric balloon system
- Sleeve gastrectomy group (Experimental): Operation way: sleeve gastrectomy
  Using the sleeve gastrectomy to treat obesity.
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Intragastric balloon system — Intragastric balloon system (PA450) developed and produced by Changzhou Zhishan Medical Technology Co., Ltd. It is a swallowable capsule intragastric balloon.The degradable material on the intragastric balloon can be degraded naturally, and the balloon is naturally discharged from the body through the gastrointestinal tract
  Arms: Intragastric balloon system group
Procedure: Sleeve gastrectomy — Sleeve gastrectomy is the use of laparoscopy to cut out the greater curvature of the stomach, mainly for weight loss.
  Arms: Sleeve gastrectomy group

SUMMARY:
This is a prospective, single-center, randomized, open-label, parallel-controlled clinical trial to compare the changes in brain function after intragastric balloon and sleeve gastrectomy.

DETAILED DESCRIPTION:
To compare the changes in brain function in obese patients after intragastric balloon and sleeve gastrectomy. This clinical trial is a prospective, single-center, randomized, open-label, parallel-controlled study. One group uses intragastric balloon system developed by Changzhou Zhishan Medical Technology Co., Ltd, and the other groups underwent sleeve gastric surgery. Before patients are enrolled in this clinical study, the researchers will do a detailed screening of the subjects based on the inclusion criteria and the exclusion criteria to determine if the patients are appropriate for the clinical study. Patients who meet the conditions of the study will be required to sign an informed consent form. They are divided into different groups according to their own wishes. To evaluate the primary outcome measures and secondary outcome measures and to observe the changes in brain function. Finally, investigators used functional MRI, questionnaire, and laboratory examination to evaluate the weight loss effect and appetite change through the comparison of the data obtained from the different groups during the treatment.

ELIGIBILITY:
Inclusion Criteria:

18 ≤ age ≤ 65, regardless of gender;

* BMI ≥ 27.5kg/m2 and ≤ 40kg / m2;
* Those who have tried other weight loss methods in the past but are not satisfied with the results;
* Willingness to comply with the study requirements, including willingness to avoid the use of drugs or other substances for weight loss during the follow-up study;
* Right handed, avoid using antibiotics and probiotics within 3 month before enrollment;
* Be able to take proton pump inhibitors and antiemetics according to the regulations of the researcher;
* It can walk completely independently without any serious chronic orthopedic diseases;
* Be willing to avoid the use of non-steroidal anti-inflammatory drugs during the study, including aspirin, diclofenac, ibuprofen, naproxen or other known gastric irritants;
* Willing to accept gastroscopy;
* Voluntarily participate in the trial and sign the informed consent form.

Exclusion Criteria:

* Patients with previous or current diagnosis of ketoacidosis;
* Symptomatic congestive heart failure, arrhythmia or unstable coronary artery disease;
* Currently suffering from respiratory diseases such as chronic obstructive pulmonary disease (COPD), pneumonia or lung cancer;
* Have undergone weight loss surgery before enrollment in the study, or may have undergone weight loss surgery during the study;
* Before the study, he used intragastric medical devices to lose weight;
* Had acute or chronic pancreatitis within 12 months before enrollment;
* Previous or current history of small bowel obstruction
* Obesity caused by genetic endocrine reasons (test results of cortical hormone and thyroid hormone, clinically significant abnormalities determined by the researcher) and not fully controlled by drugs;
* Esophageal, gastric or duodenal diseases (including hiatal hernia (≥ 2cm), paraesophageal hernia, polyps, acute erosive gastritis, cancer, varices, diverticulum, gastroparesis, ulcer, stenosis, achalasia of cardia complicated with esophagitis, etc.);
* Systemic corticosteroid anticoagulants (such as warfarin, dabigatran or antiplatelet drugs), immunosuppressive drugs (such as imidazole thiopurine, cyclosporine), prescription or over-the-counter weight loss drugs, drugs known to cause significant weight gain or weight loss, such as anesthetics, opioids or diazepines), insulin Antiepileptic drugs (such as clonazepam and phenytoin sodium), antiarrhythmic drugs (such as amiodarone); Other drugs that may cause weight change include: drugs that can significantly increase weight (such as glucocorticoids, insulin secretagogues, thiazolidinediones, atypical antipsychotics, sodium valproate, lamotrigine, antidepressants), and drugs that can significantly reduce weight (such as glucagon like peptide-1 receptor agonists α- Glucosidase inhibitor, zonisamide, topiramate, fluoxetine, bupropion, etc.);
* Night eating syndrome or bulimia;
* Unwilling to avoid any reconstruction and / or plastic surgery that may affect body weight during the study, such as mastoplasty and liposuction;
* Patients with inflammatory bowel disease (such as Crohn's disease and ulcerative colitis);
* Previous history of malignant tumor;
* Women of childbearing age whose pregnancy test is not negative before examination, lactating women, or who plan to conceive within half a year;
* Past or current drug or alcohol abuse.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Mean overall weight loss response rate | 16 weeks after operation
  (Weight loss / total weight before treatment × 100%≥5%) number of subjects / total number of subjects × 100%

SECONDARY OUTCOMES:
Mean total weight loss percentage of subjects（%TWL） | The 16th, 24th and 32nd weeks after operation
  Weight loss / total weight before treatment × 100%
Weight loss maintenance | The 16th, 24th and 32nd weeks after operation
  Weight loss and maintenance of subjects
Impact Of Weight On Quality Of Life-Lite (IWQOL-Lite) Questionnaire | The 16th, 24th and 32nd weeks after operation
  Change in obesity-specific health-related quality of life as measured by Impact Of Weight On Quality Of Life-Lite (IWQOL-Lite) Questionnaire total score from baseline to 32 weeks Minimum 0 Maximum 100 Higher score means better
Questionnaire | Preoperative and postoperative weeks 16, 24 and 32
  Evaluation of postoperative appetite related questionnaire（the Hospital Anxiety and Depression Scale, the Three-Factor Eating Questionnaire R21, the Yale Food Addiction Scale 2.0）
Gastrointestinal hormone | Preoperative and postoperative weeks 16, 24 and 32
  Changes of gastrointestinal hormone（ghrelin，leptin，cholecystokinin，adiponectin） levels after operation
Brain function | Preoperative and postoperative weeks 16, 24 and 32
  Brain functional magnetic resonance imaging
Correlation of fecal microbial profile with obesity | Preoperative and postoperative weeks 16, 24 and 32
  Analysis of fecal microbial profile using 16s rRNA sequencing

CONTACTS AND LOCATIONS:
Overall Officials: Shaihong Zhu, M.D., Principal Investigator — The Third Xiangya Hospital of Central South University
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China